CLINICAL TRIAL: NCT05574634
Title: Losing Specificity: the Role of the Locus Coeruleus in Age-related Distractibility
Brief Title: The Role of the Locus Coeruleus in Age-related Distractibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-514
Record Dates: First submitted 2022-09-13; First posted 2022-10-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Aging; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will not be aware that there are two alternate versions of the attention practice program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older adult participants (Experimental): Older adult participants in the study will complete one of two variants of an attention practice program and that will be preceded by, and followed by, an fMRI scan session featuring an attention task
  Interventions: Behavioral: Tablet based adaptive multimodal attention practice program; Behavioral: Tablet based adaptive criterion task practice program
- Younger adult participants (No Intervention): Younger adult participants in the study will complete one fMRI scan session featuring an attention task

INTERVENTIONS:
Behavioral: Tablet based adaptive multimodal attention practice program — An adaptive at-home tablet-based program that includes variants of the Flanker Task, the Stroop Task, and a Visual Tracking Task. Each session of practice will include up to ten minutes with each of these task types, and the tasks will increase in difficulty in a way that further taxes attention (such as through more distractors or more incongruent trials) as participant performance improves.
  Arms: Older adult participants
Behavioral: Tablet based adaptive criterion task practice program — An adaptive, at-home tablet-based variant of the criterion task, that is, the selective attention/distraction task used during the scanning portion of the human participant portions of the study, that takes up to 25 minutes to complete each session.
  Arms: Older adult participants

SUMMARY:
A growing body of research has highlighted the importance of frontal regions, at both the functional and structural levels, in age-related declines in attentional and cognitive processing. However, the underlying neurobiological pathophysiological changes in the brain that contribute to these declines are still largely unclear. The objective of this proposal is to investigate neural mechanisms of age-related attentional distractibility, focusing on the neural circuit initiated from the locus coeruleus (LC). In the current proposal, the investigators will test the hypothesis that the neural disconnectivity of LC with the salience network (SN) drives failures of ignoring distractors in older adults. The investigators will examine how LC-SN connectivity is associated with selective attention performance, and how improved LC-SN connectivity through a cognitive training program may lead to improved attentional performance.

ELIGIBILITY:
Inclusion:

* Healthy adult participants
* No younger than 18 and no older than 75 yrs of age
* Ability to provide written informed consent

Exclusion:

* History of surgery involving metal implants
* Possible metal fragments in the eyes
* Pacemaker
* A history of claustrophobia
* Braces
* Weighing over 250 pounds
* Pregnant or possibility of being pregnant.
* Severe medical or psychiatric conditions (e.g., blind or deaf, head trauma)
* Learning disabilities or developmental disabilities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in accuracy on the place-face selective attention task after two weeks | Scan before and after attentional practice (2 weeks between scans)
  During this task, participants will be presented to with target place stimuli overlaid on nonexpressive faces) and be asked to identify categories of place images ('building' to 'house') selectively as soon as possible while ignoring overlapped faces. The investigators will also include place only images to measure participants' baseline neural activation when there is no distractor. Each image condition will be presented in a mixed event related design that includes 15 blocks for each condition as a function of image type (overlaid vs. place-only). The block order will be counterbalanced and each block will be separated by a 10-s blank screen.
Change in fMRI LC-SN connectivity after two weeks | Scan before and after attentional practice (2 weeks between scans)
  An fMRI measure of LC-SN connectivity

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Ho Lee, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No